CLINICAL TRIAL: NCT02807675
Title: A Phase 1 Study of the Safety and Tolerability of a Single Dose Administration of CVT- 301 (Levodopa Inhalation Powder) When Administered for Early Morning OFF Symptoms in Patients With Parkinson's Disease
Brief Title: A Study of the Safety and Tolerability of a Single Dose Administration of CVT-301 (Levodopa Inhalation Powder)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acorda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVT-301-009
Record Dates: First submitted 2016-06-17; First posted 2016-06-21 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — SMG1 protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CVT-301, levodopa inhalation powder (LIP) (Experimental): designed to deliver l-dopa to the lung using the CVT-301 inhaler.
  Interventions: Drug: CVT-301, LIP
- Placebo (Placebo Comparator): Administered in the same way as the investigational product, except that it does not contain l-dopa.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CVT-301, LIP — All subjects will receive 1 dose of CVT-301 and 1 dose of placebo inhalation powder, to be taken concomitantly with their standard oral medication in 2 dosing periods. The order of treatment will be randomized, with subjects assigned to 1 of 2 sequences CVT-301 (A) administered first, followed by placebo (B), or the reverse order (BA)
  Arms: CVT-301, levodopa inhalation powder (LIP)
Other: Placebo — All subjects will receive 1 dose of CVT-301 and 1 dose of placebo inhalation powder, to be taken concomitantly with their standard oral medication in 2 dosing periods. The order of treatment will be randomized, with subjects assigned to 1 of 2 sequences CVT-301 (A) administered first, followed by placebo (B), or the reverse order (BA)
  Arms: Placebo

SUMMARY:
This study is a double-blind, randomized, placebo-controlled, 2-way crossover study to evaluate the safety of CVT-301 levodopa (l-dopa) when co- administered with the first daily dose of oral levodopa/carbidopa for early morning OFF symptoms in patients with Parkinson's disease (PD).

DETAILED DESCRIPTION:
An "OFF state" is defined as the time when medication is no longer providing benefit with respect to mobility, slowness, and stiffness. OFF episodes may be heralded by non-motor symptoms (e.g., pain, anxiety) prior to the appearance of motor symptoms.

ELIGIBILITY:
Inclusion Criteria:

* have idiopathic PD (i.e., not induced by drugs or other diseases) as defined by fulfilling Steps 1 and 2 of the United Kingdom (UK) Brain Bank criteria, diagnosed after the age of 30 years
* diagnosis of Parkinson's disease and motor fluctuations and early morning OFF symptoms
* classified as Stage 1 to 3 on the modified Hoehn and Yahr scale for staging of PD severity (in an ON state)
* subjects who are on a l-dopa-containing therapy, not including Rytary (or equivalent), must be stable on oral l-dopa-containing therapy for at least 2 weeks prior to the Screening Visit with a l-dopa/decarboxylase inhibitor (DDI)-containing regimen
* subjects who are on a l-dopa-containing therapy, when including Rytary (or equivalent), should be on a stable dose for at least 6 weeks prior to the Screening Visit
* the frequency of l-dopa administrations must be at least 3 times during the waking day and a total daily l-dopa dose of ≤ 1600 mg.
* on a stable regimen of their standard PD medications
* on a stable regimen of any blood pressure reducing medications (if applicable) for at least 30 days prior to screening
* forced expiratory volume in one second (FEV1) ≥60% of predicted for race, age, sex, and height and FEV1/FVC (forced vital capacity) ratio ≥70%
* no clinically significant abnormalities that would affect ability to complete study as determined by medical history, physical examination, electrocardiogram, clinical laboratory test results
* negative drug and alcohol testing
* negative pregnancy test for all women.

Exclusion Criteria:

* participated in any prior study with CVT-301
* dyskinesia of a severity that would significantly interfere with the subject's ability to participate or perform study procedures (as determined by the UPDRS Part 4)
* any contraindication to performing routine spirometry or who are unable to perform a spirometry maneuver
* have a current history of symptomatic orthostatic hypotension or are treated with medications to treat orthostatic hypotension (for example droxidopa, fludrocortisone), if they have severe dysautonomia
* have chronic obstructive pulmonary disease (COPD), asthma, or another chronic respiratory disease within the last 5 years.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-06; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Number of patients with Adverse Events (AEs) including Serious AEs | up to 9 days

SECONDARY OUTCOMES:
Examiner rated time to ON comparisons between treatments (CVT-301 and placebo) | day 1 and day 3
  An "ON state" is defined as the time when medication is providing benefit with respect to mobility, slowness, and stiffness, and may or may not be providing complete alleviation of all PD symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Komjathy, MD, Study Director — Acorda Therapeutics
Locations (11):
- United States (11):
  - Site #9015, Fountain Valley, California
  - Site #9002, Boca Raton, Florida
  - Site #9017, Hallandale, Florida
  - Site #9008, St. Petersburg, Florida
  - Site #9018, Sunrise, Florida
  - Site #9004, Tampa, Florida
  - Site #9016, Atlanta, Georgia
  - Site #9009, Chicago, Illinois
  - Site #9003, Farmington Hills, Michigan
  - Site #9005, West Bloomfield, Michigan
  - Site #9007, Nashville, Tennessee